CLINICAL TRIAL: NCT02492997
Title: Clinical Evaluation of Venus Versa Octipolar Applicator for Reduction of Abdomen Circumference
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was terminated early due to slow enrollment.
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS0615
Record Dates: First submitted 2015-06-19; First posted 2015-07-09 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Lipodystrophy
Keywords: body fat
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Group treated with the active Venus Versa octipolar applicator and the glycerine gel.
  Interventions: Device: Venus Versa; Other: Glycerine gel
- Control Group (Sham Comparator): Group treated with the inactive Venus Versa octipolar applicator and the glycerine gel.
  Interventions: Device: Venus Versa; Other: Glycerine gel

INTERVENTIONS:
Device: Venus Versa — The Venus Versa system is a console that supports an applicators that simultaneously emits radio frequency (RF) and a Pulsed Magnetic Field (PEMF). This combination of energy can raise the temperature of treatment area quickly and homogeneously. The Pulsed Magnetic Field is induced by short pulses of electrical current through coil in the applicator. The magnetic field penetrates into the skin and results in Foucault (Eddy) electrical currents around the cell membranes of the treated tissues. Foucault currents change the electrical potential of charged receptors on the bi-lipid cell membrane layer of dermal cells, which results in the stimulation of molecular and cellular activities and reactions.
Other: Glycerine gel — Gel used to protect the skin from the RF energy and to assist with energy distribution

SUMMARY:
The octipolar applicator is intended for circumference reduction treatment by reduction of adipose size and enhancement of collagen synthesis as the result thermal and non-thermal collagen stimulation. This trial is intended to evaluate the effect of radio frequency (RF) and pulsed electromagnetic fields (PEMF) treatment on circumference reduction.

DETAILED DESCRIPTION:
This is a multi-site, prospective, controlled, randomized, double blinded clinical trial. This study is designed to evaluate the safety and efficacy of a series of treatments using the Venus Versa Octipolar applicator. Up to 60 healthy subjects at 10 sites shall be recruited by the investigator from within the investigator's subject population. Subjects shall have abdomen circumference to reduce for the designated treatment area.

Each subject will undergo 6 treatments at an interval of one treatment per week for six consecutive weeks. There will be a one month follow up which will occur 4 weeks after the 6th treatment.

At the first treatment visit, the investigator will collect demographic and medical information and randomization will take place. Subjects have an equal opportunity to be selected for the treatment or the control group.

The duration of the treatment session will be approximately 60 minutes. Expected immediate response includes temporary mild to moderate erythema and/or edema. Skin safety assessments will be conducted by the investigator after each treatment session and at the follow-up visit.

Photography will be conducted at baseline, the beginning of 4th & 6th treatment and at 1 month follow up visit. Subjects will be asked to complete a questionnaire after each treatment and at the one month follow up visit.

Circumference measurements will be conducted at base line, before each treatment and at follow up visit. The treatment will be considered successful if the treated area circumference, reduces by at least 2.5 cm.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) score is greater than 18.5 and less than 29.9 - normal to overweight, but not obese.
* Willingness to refrain from a change in diet/drinking/exercise/medication regimen for the entire course of the study.
* For female of child bearing potential - using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, Intra Uterine Device (IUD), contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant or planning to become pregnant, having given birth less than 9 months ago, and/or breastfeeding.
* Having any active electrical implant anywhere in the body,
* Having a permanent implant in the treated areas
* Having received treatment with laser, RF or other devices in the treated areas within 6 months of treatment or during the study.
* Having undergone a liposuction surgery or any contouring treatment in the areas intended for treatment within 2 years of treatment
* Having or undergoing any form of cancer
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders.
* Having a anticoagulative or thromboembolic condition or taking anticoagulation medications
* History of immunosuppression/immune deficiency disorders
* Suffering from hormonal imbalance which may affect weight or cellulite
* History of significant lymphatic drainage problems.
* History of keloid scarring or of abnormal wound healing.
* History of being especially prone to bruising.
* History of epidermal or dermal disorders
* Use of isotretinoin within 6 months
* Significant change in diet or exercise regimen within a month of enrollment or during this study and/or weight loss or gain of 10 lbs (4.5 kgs) within 2 months of enrollment or during this study.
* Participation in a study of another device or drug within 1 month prior to enrollment or during this study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Mancuso, Study Director — Venus Concept
Locations (1):
- J Dermatology and Allergy, Fort Lee, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was opened in March 2015. By time of study closure in October 106, only 44 of the planned 60 subjects had been enrolled to the study. As such, the trial was terminated due to slow enrollment.
Pre-assignment Details: Two subjects were reported to have been screen failed.
Groups:
- Treatment Group: Group treated with the active Venus Versa octipolar applicator and the glycerin gel.
  Venus Versa: The Venus Versa system is a console that supports an applicators that simultaneously emits radio frequency (RF) and a Pulsed Magnetic Field (PEMF). This combination of energy can raise the temperature of treatment area quickly and homogeneously. The Pulsed Magnetic Field is induced by short pulses of electrical current through coil in the applicator. The magnetic field penetrates into the skin and results in Foucault (Eddy) electrical currents around the cell membranes of the treated tissues. Foucault currents change the electrical potential of charged receptors on the bi-lipid cell membrane layer of dermal cells, which results in the stimulation of molecular and cellular activities and reactions.
  Glycerine gel: Gel used to protect the skin from the RF energy and to assist with energy distribution
- Control Group: Group treated with the inactive Venus Versa octipolar applicator and the glycerin gel.
  Venus Versa: The Venus Versa system is a console that supports an applicators that simultaneously emits radio frequency (RF) and a Pulsed Magnetic Field (PEMF). This combination of energy can raise the temperature of treatment area quickly and homogeneously. The Pulsed Magnetic Field is induced by short pulses of electrical current through coil in the applicator. The magnetic field penetrates into the skin and results in Foucault (Eddy) electrical currents around the cell membranes of the treated tissues. Foucault currents change the electrical potential of charged receptors on the bi-lipid cell membrane layer of dermal cells, which results in the stimulation of molecular and cellular activities and reactions.
  Glycerine gel: Gel used to protect the skin from the RF energy and to assist with energy distribution
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Gained Weight | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Group treated with the active Venus Versa octipolar applicator and the glycerin gel.
- Control Group: Group treated with the inactive Venus Versa octipolar applicator and the glycerin gel.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
Abdominal circumference [Mean (Standard Deviation); unit: cm] — Abdominal circumference measurement (cm) from at a height from floor to abdominal umbilicus (reference point) while standing barefoot. The abdomen is measured (with a controlled tape measure) in the reference point with tape snug but not too tight. Population: Thirty-nine subjects signed consent. Only thirty CRFs were returned to sponsor on closure of study. Remaining nine CRFs were assumed to be lost.
  cm
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 91.47 (9.35) | 86.66 (8.22) | 90.74 (9.49)

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Circumference
Description: Abdominal circumference measurement of the treated area at 1 month after the last treatment performed by controlled tape measurement
Time Frame: 1 month post treatment series
Population: Of the thirty subjects who started the study, one of the treatment group and two from the control group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 14 | 13
cm | 90.18 (7.16) | 88.05 (8.78)

2. Secondary Outcome: Subject Satisfaction With Treatment
Description: Subject 5-point Likert Satisfaction Assessment Scale where 4 = Very satisfied; 3 = Satisfied; 2 = Having no opinion; 1 = Unsatisfied and 0 = Very unsatisfied.
Time Frame: 1 month post treatment series
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 14 | 13
Participants
  Very satisfied | 3 | 0
  Satisfied | 8 | 1
  Having no opinion | 2 | 5
  Unsatisfied | 1 | 3
  Very unsatisfied | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year, 7 months and 10 days.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
The trial commenced March 14, 2015 and was closed on October 25, 2016. The trial was terminated early due to insufficient recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No